CLINICAL TRIAL: NCT05309330
Title: Assessment of Symptom Patterns in Celiac Disease: A Prospective Longitudinal Survey
Brief Title: Virtual Celiac Symptoms Study in Adults and Teenagers
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-101-5001
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Signs and Symptoms; Digestive; Quality of Life; Diet; Gluten-Free
MeSH Terms: conditions — Celiac Disease; Signs and Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with CeD: Participants diagnosed with CeD will be observed prospectively for CeD symptom patterns over a 3-month period.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The goal of this study is to better understand the symptoms and impacts of celiac disease (CeD). Participants use a smart phone online app to answer daily questionnaires about symptoms and life with CeD for 12 weeks. There are no blood draws, gluten challenges, medications, or doctor visits required.

DETAILED DESCRIPTION:
This is an observational, prospective study to measure symptoms and impacts of CeD.

This study will assess CeD symptom patterns over a 3-month observation period. The study will enroll approximately 400 participants.

The data will be prospectively collected, via a self-reported ePRO platform accessible by smartphone.

This virtual study will be conducted in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. At least 12 years of age or older.
2. Diagnosed with CeD for at least 1 year.
3. For participants diagnosed over the age of 18: Biopsy confirmed diagnosis with CeD (participant reported).
4. For participants diagnosed under the age of 18: Blood test or biopsy confirmed diagnosis with CeD (participant reported).
5. Currently following a gluten free diet (GFD) for at least 6 months.
6. Has experienced symptoms believed by the participant to be CeD related in the last 3 months.
7. Has daily access to a smartphone as well as internet/Wi-Fi/cellular data.
8. Speaks and reads English.
9. Lives in the US (participant reported).

Exclusion Criteria:

1. Currently involved or planning to be involved in any clinical studies with an investigational drug, surgical procedure, or gluten challenge over the 3-month observation period.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants diagnosed with CeD in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Each Gastrointestinal Symptom and Tiredness Assessed by the Celiac Disease Symptom Diary (CDSD) | Up to 12 weeks
  The CDSD is a celiac specific symptom assessment tool administered daily. The symptoms measured will include diarrhea, abdominal pain, bloating, nausea/vomiting, number of bowel movements and tiredness. Presence and count of each symptom will be reported for the overall sample as well as separately for adults (age greater than or equal to [>=] 18) and adolescents (age >=12 less than [<] 18).
Number of Participants With Presence of Non-gastrointestinal (GI) Symptoms | Up to 12 weeks
  Non-GI symptoms include: Headache, Brain fog (feeling confused or disorganized, or finding it hard to put thoughts into words), Dermatitis herpetiformis (DH) or other rash (suspected to be related to gluten exposure), Joint/body pain (suspected to be related to gluten exposure), Irritability (feeling easily upset or frustrated), Mouth sores/canker sores, and others. Presence/count of each symptom will be assessed overall and separately for adults (age >=18) and adolescents (age >=12 and <18).

SECONDARY OUTCOMES:
Number of Participants With Presence/Absence of Known and Suspected Gluten Exposure | Up to 12 weeks
  This will be assessed overall and separately for adults (age >=18) and adolescents (age >=12 and <18).
Quality of Life (QoL) as Measured by the 12-Item Short Form Survey (SF-12) Version 2 (v2) | Up to 12 weeks
  QoL will be measured using SF-12v2. SF-12 is a 12-item self-report that assesses the impact of health on an individual's everyday life. Average SF-12 scores will be reported for the overall sample as well as separately for adults (age >=18) and adolescents (age >=12 and <18).
Number of Participants With Healthcare Resource Utilization (HCRU) | Up to 12 weeks
  Participants reporting the number of hospitalizations, emergency room (ER) visits, and outpatient/urgent care visits they had in the previous week. HCRU will be reported for the overall sample as well as separately for adults (age >=18) and adolescents (age >=12 and <18).
Work Productivity Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire | Up to 12 weeks
  WPAI measures the effect of general health and symptom severity on work/schoolwork productivity and regular activities during the past seven days. Average WPAI scores will be reported for the overall sample as well as separately for adults (age >=18) and adolescents (age >=12 and <18).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda, Lexington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/f79a24e4008a4981?idFilter=%5B%22TAK-101-5001%22%5D